CLINICAL TRIAL: NCT01498146
Title: Stroke Prior to Diagnosis of Atrial Fibrillation Using Longterm Observation With Implantable Cardiac Monitoring Apparatus Reveal(SURPRISE) -the SURPRISE Study
Brief Title: Finding Atrial Fibrillation in Patients With Unexplained Stroke Using Longterm Cardiac Monitoring
Acronym: SURPRISE
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Associate Research Professor, Consultant neurologist, Bispebjerg Hospital
Other Study IDs: H-4-2010-014
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Stroke
Keywords: cryptogenic stroke; atrial fibrillation; longterm monitoring; loop recorder
MeSH Terms: conditions — Stroke; Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The SURPRISE study investigates atrial fibrillation(AFIB) in patients with a previous unexplained stroke. It uses long term monitoring of the heart of up to three years, searching for paroxysmal atrial fibrillation(PAF) otherwise undetected in this population.

DETAILED DESCRIPTION:
The SURPRISE study investigates the patients with cryptogenic stroke or transient ischemic attack (TIA), monitoring them with a cardiac loop recorder for up to three years.

it aims at estimating the amount of paroxysmal atrial fibrillation within our population of cryptogenic stroke patients.

Standard workup for a stroke patient does offer cardiac evaluation, but monitoring is limited to the time admitted, often just a few days.

ELIGIBILITY:
Inclusion Criteria:

* Computerized Tomography (CT) or Magnetic resonance imaging (MRI) verified cryptogenic stroke or TIA;
* > 18 years of age,
* the ability to provide a written consent

Exclusion Criteria:

* prior or known AFIB
* AF found during work up including 24 hour telemetric monitoring.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the patients are included from the investigators stroke unit and day clinic
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, MD, PhD, DMSci, Principal Investigator — University of Copenhagen
Locations (1):
- Bispebjerg Hospital, University Hospital of Copenhagen, dept of Neurology, Copenhagen, Denmark

REFERENCES:
- [Derived] Biering-Sorensen T, Christensen LM, Krieger DW, Mogelvang R, Jensen JS, Hojberg S, Host N, Karlsen FM, Christensen H. LA emptying fraction improves diagnosis of paroxysmal AF after cryptogenic ischemic stroke: results from the SURPRISE study. JACC Cardiovasc Imaging. 2014 Sep;7(9):962-3. doi: 10.1016/j.jcmg.2014.02.003. Epub 2014 Apr 9. No abstract available. PMID 24726253